CLINICAL TRIAL: NCT03143946
Title: Towards Optimal Personalized Diet and Vitamin Supplementation in Patients With a Neuroendocrine Tumor
Brief Title: DIVIT Study Diet and Vitamin Supplementation in Patients With a Neuroendocrine Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201600626
Record Dates: First submitted 2016-10-11; First posted 2017-05-08 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumor
Keywords: neuroendocrine tumor; vitamin; diet
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin supplement and diet advice (Experimental): Single arm. Patient be prescribed vitamin supplement if vitamin deficiencies are diagnosed and will get diet advice
  Interventions: Dietary Supplement: Vitamin supplement;; Other: Diet advice

INTERVENTIONS:
Dietary Supplement: Vitamin supplement; — Vitamin K, vitamin A, vitamin D, vitamin E, nicotinamide, vitamin B12
Other: Diet advice

SUMMARY:
This study aims to investigate if the proportion of neuroendocrine tumor (NET) patients with normal vitamin values can be increased, with vitamin suppletion and a personalized diet, Effects of the intervention will be evaluated by quantitative analysis of blood and urine and questionnaires. The measurements, will be performed at baseline (t=0), after 4 weeks (t=4) and after 18 weeks at end of study (t=18). Furthermore at t=18 a semi-qualitative interview will be performed.

DETAILED DESCRIPTION:
Objective:

This study aims to investigate if the proportion of NET patients with normal vitamin values can be increased, with vitamin suppletion and a personalized diet.

Methods:

This is a single center 18-week open-label, non-comparative, single-arm, intervention study. After inclusion and the first measurements, adult patients with metastasized or irresectable NET will continue with four weeks of standard treatment. After these four weeks participants with vitamin values below normal will get vitamin suppletion for each deficient vitamin and all participants will get the dietary intervention during 14 weeks. Effects of the intervention will be evaluated by quantitative analysis of blood and urine and questionnaires. The measurements, including; baseline characteristics, quantitative analysis of blood and urine and questionnaires will be performed at baseline (t=0), after 4 weeks (t=4) and after 18 weeks at end of study (t=18). Furthermore at t=18 a semi-qualitative interview will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18 years
* NET-patients with serotonin producing or non-serotonin producing tumors, with gastro-intestinal, pancreatic, bronchopulmonary or unknown primary tumor site and with metastasized or irresectable disease
* Ability to comprehend Dutch (both reading and writing).
* Written informed consent provided.
* Use of somatostatin analogue for > 6 months.

Exclusion Criteria:

* Estimated life expectancy less than 6 months.
* Patients who have a history of another primary malignancy, except for radical and adequately treated malignancies from which the patient has been disease free for ≥ 1 year.
* Major abdominal surgery during study period.
* Patients already participated in the DIVIT-pilot study
* Known hypersensitivity of (components of) somatostatin analogue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
the change in the proportion of patients with normal vitamin values | 18 weeks
  the change in the proportion of patients with normal vitamin values measured with quantitative analysis of blood and urine

SECONDARY OUTCOMES:
nutrition state | 18 weeks
  As measured with the total score with Patient-Generated Subjective Global Assessment (PG/SGA).
distress | 18 weeks
  measured by the distress thermometer and problem list
problems | 18 weeks
  as measured with the problem list.(the mean of each item)
change in quality of life | 18 weeks
  determined by the QLQ-GINET21 (a NET-specific EORTC quality of life questionnaire) and the cancer-specific EORTC QLQ-C30,
difference in the self-reported healthy eating pattern. | 18 weeks
  as measured with a self-constructed scale

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek ME Walenkamp, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No